CLINICAL TRIAL: NCT02275689
Title: Alternative Treatment of Rotator Cuff Tendinopathy
Brief Title: Radiofrequency Microtenotomy for Treatment of Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/1133
Record Dates: First submitted 2014-10-22; First posted 2014-10-27 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2016-12

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Rotator cuff; Tendinosis; Impingement; radiofrequency
MeSH Terms: conditions — Shoulder Impingement Syndrome; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arthrocopic acromioplasty (Active Comparator): Surgical intervention with arthroscopic acromioplasty, bursectomy and subacromial decompression
  Interventions: Procedure: Arthroscopic acromioplasty
- Radiofrequency microtenotomy (Active Comparator): Surgical intervention With arthroscopic radiofrequency microtenotomy
  Interventions: Procedure: Microtenotomy
- Physical therapy (No Intervention): Muscle strength training, home trainings programme

INTERVENTIONS:
Procedure: Arthroscopic acromioplasty — Surgical intervention With arthroscopic acromion resection
  Arms: Arthrocopic acromioplasty
Procedure: Microtenotomy — Arthroscopic radiofrequency microtenotomy of rotator cuff tendon
  Arms: Radiofrequency microtenotomy

SUMMARY:
This study compare the outcome (pain, function) after Radiofrequency microtenotomy (group I) and acromioplasty (group II) for treatment of rotator cuff tendinosis in the shoulder.

The outcome of both methods will be compared to the physical therapy treatment (groupIII)

DETAILED DESCRIPTION:
Rotator cuff tendinosis cause pain and disability of the shoulder. Tendinosis, sometimes complicated by partial rupture, appears to be the major lesion in chronic rotator cuff tendinopathy. Important features is a poor intrinsic ability to heal.

Several patients receive treatment for shoulder tendinosis each year. Conservative treatments options include rest, stretching, strengthening, ice and/or physical therapy are used with difference results. A traditional surgical treatments (acromioplasty) have been reported with variable results..

The aim of this study is to evaluate improvement of VAS and functionality using Constant score before and after treatment of rotator cuff tendinosis using radiofrequency-plasma based microtenotomy in comparison to traditional acromioplasty and physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Impingement pain in the shoulder at least 3 months
* MRI of shoulder reveal tendinosis
* Classification of Acromion morphology by RTG and or MRI
* daily pain

Exclusion Criteria:

* inflammatory joint disease
* Other comorbidity in the shoulder as instability, osteoarthritis or rotator cuff tear
* serious illness

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in VAS for pain | every 2 weeks. during 6 months
  The patients will have a clinical control 6,12 weeks and 6 months postoperatively. The VAS will be registered every 2 weeks via SMS during 6 months
Change from baseline in VAS for pain, | 6 weeks, 6 months, and 12 months

SECONDARY OUTCOMES:
Change from baseline in functionality measured by constant score | 6 weeks, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Meknas, MD, PhD, Principal Investigator — University Hospital of North Norway. 9038-Tromsø. Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway